CLINICAL TRIAL: NCT06733454
Title: Remote EEG Experiences With Families
Brief Title: REEF: Remote EEG Experiences With Families
Acronym: REEF
Status: Enrolling by invitation | Type: Observational
Sponsor: New York University (Other)
Responsible Party: Sponsor
Other Study IDs: NYU-IRB-FY2024-9108
Record Dates: First submitted 2024-12-09; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Healthy
Keywords: Pediatric EEG

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
The goal of this observational study is to learn about the usability of portable EEG sensors (REMI) in the home with infants and young children. The main question it aims to answer is: Can families comfortably use portable EEG sensors (REMI) in the home with their children? Families will wear the REMI sensors for an extended period of time (30 minutes to 1 week) and answer online survey questions.

DETAILED DESCRIPTION:
There has been significant innovation in remote testing procedures over the past few years, accelerated in part as a result of the COVID-19 pandemic-related testing restrictions. Shifts to remote testing have included standardization of methods for survey administration and adaptations of traditional in-lab paradigms for use in remote assessments. The current project will develop and standardize a remote protocol measuring infant brain function using wireless, portable, user-friendly, single-channel EEG sensors. Infant cortical activity will be collected using the REMI (Remote EEG Monitoring System), a wireless, single-channel sensor. The sensors are applied to the head using specially designed infant-friendly adhesive stickers (to avoid skin irritation). Families of children between the ages of 1 month and 24 months will be eligible to participate in this study. Experimenters will initiate the sensors and will instruct families on how to use the REMI system independently (i.e., changing adhesive stickers when necessary). Families will then record child EEG for an extended period of time (30 minutes to 2 weeks). When recording is complete, the family will mail back all equipment to the lab.

ELIGIBILITY:
Inclusion Criteria:

* Child is between the ages of 1 month and 24 months of age

Exclusion Criteria:

* Child has known neurodevelopment disorder
* Legal guardian is under 18 years of age

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Families with children 1-month to 24-months of age will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants who independently recorded at least 30 minutes of data | Up to 2 weeks
  Examine the length of time for each recording as well as qualitative information on feasibility

CONTACTS AND LOCATIONS:
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No